CLINICAL TRIAL: NCT00166790
Title: Detection of Minimal Amount of Human Chorionic Gonadotropin by Interferometry in Gestational Trophoblastic Disease
Brief Title: Detection of Human Chorionic Gonadotropin by Interferometry in Gestational Trophoblastic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 9461700666; NSC 94-2314-B-002-221
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Trophoblastic Neoplasms
Keywords: Human Chorionic Gonadotropin; Dual Polarization Interferometry,; Gestational Trophoblastic Neoplasms
MeSH Terms: conditions — Trophoblastic Neoplasms; Gestational Trophoblastic Disease | interventions — Vacuum Curettage

INTERVENTIONS:
Drug: chemotherapy agents
Procedure: suction curettage

SUMMARY:
We will try to use the novel analytical technique -Dual Polarisation Interferometry (DPI),to achieve detection the minimal amount of the human chorionic gonadotropin for early detection and strict monitor of the GTD.

DETAILED DESCRIPTION:
1 Gestational trophoblastic disease (GTD) consists of a spectrum of disorders that are characterized by an abnormal proliferation of trophoblastic tissue. They include hydatidiform mole, invasive mole, choriocarcinoma and placental site trophoblastic tumor (PSTT). The incidence of molar pregnancies in Asian countries is 7 to 10 times greater than the reported incidence in Europe or North America. Although previously a lethal disease, GTD is considered today the most curable gynecologic cancer. This progress can be attributed to an available tumor markerhuman chorionic gonadotropin (hCG), chemosensitivity, and the incorporation of aggressive multimodality therapy. However, a delay in the diagnosis may increase the patient's risk of developing malignant GTN and adversely affect response to treatment, and therefore the prompt identification of GTN is important. Approximately 20% of patients will develop malignant sequelae requiring administration of chemotherapy after evacuation of hydatidiform moles. The overall cure rate for patients with nonmetastatic disease and low-risk metastatic disease is nearly 100% .When chemotherapy is given for an additional 1-2 cycles after the first normal hCG value, recurrence rates are less than 5%. In contrast, in high risk metastatic disease, chemotherapy is continued until hCG values have normalized, followed by at least two or three courses of maintenance chemotherapy in the hopes of eradicating all viable tumors. Despite the use of sensitive hCG assays and maintenance chemotherapy, up to 13% of patients with high-risk disease will develop recurrence after achieving an initial remission. Conventionally, serial quantitative serum hCG determinations should be performed using commercially available assays capable of detecting β-hCG to baseline values(<5 mIU/ml). However, the amount of hCG produced correlates with tumor volume so that a serum hCG of 5 mIU/mL corresponds to approximately 104 to 105 viable tumor cells. Therefore, detection of minimal amount of human chorionic gonadotropin (<5 mIU/ml) is crucial, it could help to early detect the GTD and strictly monitor the residual activity of the tumor after chemotherapy.

Dual Polarisation Interferometry (DPI) is an analytical technique used to understand the real-time structure and behaviour of a wide range of molecular systems and interactions through quantitative measurement including molecular size, density and mass. DPI has been successful across a range of applications, including proteins,lipids, nucleic acids, lectins, surfactants, polymers, interfacial studies, surface characterisation and nanotechnology.

Herein, we are trying to use the novel analytical technique -Dual Polarisation Interferometry (DPI),to achieve detection the minimal amount of the human chorionic gonadotropin for early detection and strict monitor of the GTD. Under this circumstance, maintenance chemotherapy is continued until hCG values is totally undetectable, in the hopes of eradicating all viable tumors. Besides this method could be more precise in sensitivity and specificity to avoid the false positive result which could led to unnecessary chemotherapy or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Hydatidiform Mole
* Choriocarcinoma
* Gestational Trophoblastic Neoplasms

Exclusion Criteria:

* Unwilling to participate in the study

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: GTD
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
HCG LEVEL | REMISSION

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Jien Chen, MD, PhD, Principal Investigator — National Taiwan university Hospital, Department of Obstetrics and Gynecology
Locations (1):
- National Taiwan University Hospital Department of Obstetrics and Gynecology, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Lichtenberg ES. Gestational trophoblastic tumor after medical abortion. Obstet Gynecol. 2003 May;101(5 Pt 2):1137-9. doi: 10.1016/s0029-7844(03)00062-0. PMID 12738129
- [Background] Behtash N, Ghaemmaghami F, Honar H, Riazi K, Nori A, Modares M, Mousavi A. Is normal beta-hCG regression curve helpful in the diagnosis of persistent trophoblastic disease? Int J Gynecol Cancer. 2004 Sep-Oct;14(5):980-3. doi: 10.1111/j.1048-891X.2004.14538.x. PMID 15361212